CLINICAL TRIAL: NCT02565641
Title: An Open-label, Phase II Study of Capecitabine Plus Gemcitabine in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: A Study of Capecitabine (Xeloda) in Participants With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML16832
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Gemcitabine

ARMS (1):
- Capecitabine + Gemcitabine (Experimental): Participants will receive oral capecitabine (830 milligrams per meter-squared [mg/m^2]) twice daily (BID) as intermittent treatment (Days 1 to 21 every 4 weeks [q4w]) along with IV infusion of gemcitabine (1000 mg/m^2) once weekly as intermittent treatment (4-week cycles of 3-week treatment period and 1-week rest period).
  Interventions: Drug: Capecitabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered orally at 830 mg/m^2 BID (equivalent to a total daily dose of 1660 mg/m^2) as intermittent treatment (given days 1 to 21 q4w).
  Other Names: Xeloda
Drug: Gemcitabine — Gemcitabine will be administered at a dose of 1000 mg/m^2 once weekly via IV infusion as intermittent treatment (repeated 4-week cycles of 3 weeks treatment and 1 week rest).

SUMMARY:
This study will evaluate the efficacy and safety of oral capecitabine plus intravenous (IV) gemcitabine in participants with locally advanced or metastatic pancreatic cancer. The anticipated time on study treatment is 3 to 12 months, and the target sample size is 56 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18 to 75 years of age
* Locally advanced or metastatic pancreatic cancer

Exclusion Criteria:

- Prior chemotherapy for pancreatic cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Overall objective response rate | At the end of 6 cycles (24 weeks)

SECONDARY OUTCOMES:
Duration of response | Up to approximately 3.5 years
Time to disease progression | Up to approximately 3.5 years
Time to response | Up to approximately 3.5 years
Time to treatment failure | Up to approximately 3.5 years
Overall survival | Up to approximately 3.5 years
Incidence of adverse events | Up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials — Hoffmann-La Roche
Locations (3):
- South Korea (3):
  - Buchun
  - Daegu
  - Seoul